CLINICAL TRIAL: NCT05998382
Title: The Effect of Parent-Mediated Intervention Program on Children's Autism Symptoms, Behavioral Problems and Parents' Stress Level in Children With Autism Spectrum Disorder Exposed to Earthquake in Turkey in February 2023
Brief Title: The Effect of Parent Mediated Intervention Program on Children With ASD Exposed to Earthquake in Turkey in February 2023
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sabri Hergüner (Other)
Responsible Party: Sponsor-Investigator, Sabri Hergüner, associate professor, Herguner Therapy Private Clinic
Organization: Herguner Therapy Private Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: February2023earthquakeinTurkey
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder; Earthquake; Behavior Problem of Childhood and Adolescence
Keywords: Autism spectrum disorder;; Social communication; Behavior Problem; Parent mediated intervention; earthquake; parental stress
MeSH Terms: conditions — Autism Spectrum Disorder; Communication; Mental Disorders

STUDY DESIGN:
Intervention Model Description: It will be realized with the participation of 24-72 months old children with autism spectrum disorder and their parents who were exposed to earthquake. The program will be announced via social media. After the applicants are evaluated, the families who will participate in the program will be given detailed information about the study and informed consent will be obtained. Before the training begins, families will be asked to fill out the Sociodemographic Data Form, Social Communication Checklist-Revised-Preschool Turkish Version, Depression Anxiety Stress Scale, ½-5 years old Child Behavior Checklist. Families will participate in the training program that will last 6 weeks. At the end of the 6th week, families will be asked to fill in the Social Communication Checklist-Revised-Preschool Turkish Version, Depression Anxiety Stress Scale, ½-5 years old Child Behavior Checklist Scale again. The change from time t1-baseline to time t2-6 weeks later was calculated by arithmetic method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): There is only one group in the study. This group will participate in a 6-week online group-based parent-mediated intervention program.
  Interventions: Behavioral: Online group-based parent-mediated intervention program

INTERVENTIONS:
Behavioral: Online group-based parent-mediated intervention program — The program is an online group-based parent-mediated intervention program implemented in 2 sessions of 2 hours once a week for 6 weeks. In the first part of the weekly sessions, the topic of that week is explained to the parents. In the second part, videos recorded by the parents are watched and feedback is given to the parents. At the end of the session, written materials about that week's practices and homework are sent to the parents

SUMMARY:
After devastating natural events such as earthquakes, individuals with special needs experience much more difficulties. There is a limited number of studies investigating the impact of disasters on individuals with autism. Studies show that resilience and recovery of pre-disaster functioning in young people with autism largely depends on their immediate inclusion in routine, intensive rehabilitation programs and the stabilization of daily life routines as much as possible. Children with autism had to interrupt their education due to many reasons such as the destruction of special education centers due to the earthquake and the temporary or permanent relocation of families to different cities. The fact that individuals with autism stayed away from education after the earthquake caused parents' stress and anxiety levels to increase. Parent involvement, a standard intervention practice in ASD, shows that teaching intervention strategies to parents can improve children's outcomes and increase parental effectiveness. Researchers aim in this study is to investigate the effect of the online group-based parent-mediated intervention program on autism symptoms, the effect on behavioral problems and the effect on parental mental health of children with autism spectrum disorder whose education life was interrupted 8 months after the earthquake, who had major changes in their lives (such as loss of relatives, loss of health, work, home, anxiety, having to change cities ...).

Online group-based intervention program ist designed to improve the interaction, play, speech and learning skills of children with autism symptoms, taking into account the earthquake conditions.

DETAILED DESCRIPTION:
Earthquakes are considered to be destructive, uncontrollable natural disasters that cause the most migration and threaten life the most. After the earthquake that occurred in L'Aquila, the capital of Abruzzo region of Italy on April 2009, children and adolescents with autism who were and were not exposed to the earthquake were followed up for 1 year in terms of adaptation skills. It was observed that adaptive skills (communication, daily living skills, socialization and motor skills) were clinically and statistically decreased one month after the earthquake in individuals with autism exposed to the earthquake. Compared to the unexposed group, adaptive skills were also found to be significantly lower. It was found that adaptation skills were 30% lower in the 6th month of the earthquake compared to the beginning and 15% lower in the 1st year.

Studies show that the recovery of resilience and pre-disaster functions in young people with autism largely depends on their immediate inclusion in routine, intensive rehabilitation programs and fixation of daily life routines as much as possible. However, after the February 06, 2023 Kahramanmaraş earthquake, many rehabilitation centers where individuals with autism received special education support were destroyed. This has made it difficult for individuals with autism to access special education support. What we know about the impact of trauma in children is that the response to traumatic events is mediated by caregivers and important people in the child's life. The fact that individuals with autism stayed away from education after the earthquake may cause parents' stress and anxiety levels to increase and their ability to cope with trauma to be negatively affected, which may naturally cause individuals with autism to be more affected by trauma.

Parental involvement in intervention in Autism Spectrum Disorder (ASD) is a standard intervention practice and research shows that teaching parents intervention strategies can improve children's outcomes and increase parental effectiveness. Parent-mediated interventions that are naturalistic, developmental and behavioral are effective in improving social and communication skills for children with ASD.

Learning that their child has ASD causes serious stress on families from the moment the diagnosis is made. High levels of parental stress have been shown to negatively affect the effectiveness of parent-mediated interventions (possibly due to interference with parental learning). Therefore, it is important to determine intervention strategies by considering parental stress in parent-mediated intervention programs.

One of the challenges for parents and children with ASD is the limited access to education, the costly nature of the education process, and sometimes the inability to make the necessary arrangements for the family to benefit from education (such as caring for other children, arranging work schedules). Online group-based trainings make it easier for families to overcome these challenges. They can access education from their own homes, it is much more cost-effective and it can be easier to make environmental arrangements. Group-based training can also help families to support and learn from each other.

The parent training program to be implemented is an online group-based intervention program implemented by parents to improve the interaction, play, speech and learning skills of children with autism symptoms. Through this program, families will be able to overcome the time, place and economic difficulties that prevent them from accessing education, and since it is a program implemented by parents, they will have the opportunity to apply it to children in a natural environment throughout the day. It will also partially prevent families from being away from education due to the destruction of education centers, relocation of educators to different cities or inaccessibility due to reasons such as death. There are a limited number of studies on the processes of readjustment of children with Autism Spectrum Disorder to daily life after natural disasters such as earthquakes that cause serious losses. There is no study on this theme conducted in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of autism must be made by a specialist
* Being in the age range of 24-72 months
* Living in one of the 10 provinces where the earthquake was felt intensely during the earthquake

Exclusion Criteria:

* Having a genetic disease

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change in autism symptom severity | baseline and 6 weeks
  Researcher examined the effect of intervention on autism symptom severity by using the change in Social Communication Checklist-Revised (SCC-R) scores. After the intervention program, whether there were significant changes in the total scores and subscales of Social Communication Checklist-Revised (SCC-R) was determined by the paired t test if it met the normal distribution conditions, and the Wilcoxon test if it did not meet the normal distribution conditions.Social Communication Checklist-Revised (SCC-R): The SCC-R is a 70-item checklist.They are summed for domain scores and a Total Score. Respondents indicate whether a child uses each skill, "Rarely/Not Yet (1)," "Sometimes, but not consistently (2)," or "Usually, at least 75% of the time (3)". The total score would then be between 70 and 215. An increase in the Total Score means that social communication skills have increased.
change in behavior problems | baseline and 6 weeks
  Researcher examined the effect of intervention on behaviour problems by using the change in 1/2-5 age Child Behavior Checklist- 1/2-5 CBCL) scores. After the intervention program, whether there were significant changes in the total scores and subscales of 1/2-5 Child Behavior Checklist was determined by the paired t test if it met the normal distribution conditions, and the Wilcoxon test if it did not meet the normal distribution conditions. 1/2-5 Child Behavior Checklist: CBCL 1.5-5 is a 99-item. The item is marked as 0 if the child does not have it, 1 if it is sometimes or somewhat true for the child, and 2 if it is very true or often true. An increase in total score means that behaviour problems is exacerbated.
change in parental stress level | baseline and 6 weeks
  It was measured by the change in the Depression Anxiety Stress Scale After the intervention program, whether there were significant changes in the total scores and subscales of Depression Anxiety Stress Scale (DASS-21) was determined by the paired t test if it met the normal distribution conditions, and the Wilcoxon test if it did not meet the normal distribution conditions.DASS-21 contains 21 items and has 3 subscales: depression, stress and anxiety. It is a Likert-type scale. As the total score increases, the severity of depression, stress and anxiety increases.

CONTACTS AND LOCATIONS:
Overall Officials: Sabri Hergüner, Assoc., Study Director — Hergüner Therapy Privat Clinic
Locations (1):
- Hergüner Therapy Private Clinic, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data can be shared 6 months after the study is publish
Access Criteria: Assoc. Prof. Dr. Sabri Hergüner will review the requests.